CLINICAL TRIAL: NCT03060746
Title: Helicobacter Pylori Sample Collection Protocol PRE-THERAPY
Brief Title: Helicobacter Pylori Sample Collection Protocol Pre Therapy Subjects
Status: Completed | Type: Observational
Sponsor: DiaSorin Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: PRE-TREAT A001
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infection; Gastric Ulcer; Nausea; Abdominal Pain; Weight Loss; Stomach Ulcer; Loss of Appetite; Bloating
MeSH Terms: conditions — Stomach Ulcer; Nausea; Abdominal Pain; Weight Loss; Anorexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Newly Diagnosed — Gastric biopsy tested by composite reference method (CRM) (histology, urease, culture) and stool sample

SUMMARY:
The primary objective is to obtain stool samples from pre-therapy subjects already undergoing evaluation for an H. pylori infection by upper esophagogastroduodenoscopy (EGD) and gastric biopsy.

DETAILED DESCRIPTION:
Stools will be collected and tested, at a later date, in a clinical performance study with an investigational H. pylori antigen assay. This study will be coordinated by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 22 years, either gender
* Subject is symptomatic showing signs and symptoms of gastritis
* Subject is not under evaluation for post-therapy follow up diagnosis
* Subject is already undergoing upper EGD and obtaining a gastric biopsy as part of routine care for H. pylori diagnosing
* Biopsy is obtained from antrum and/or corpus and is tested by CRM
* At least two of the three CRM tests are performed
* Subject whose EGD with biopsy procedure occurred ≤ 7 days prior to stool collection
* Willing and able to sign the IRB approved Informed Consent form for this project, or able to provide Informed Consent in accordance with 21 CFR 50 Subpart B

Exclusion Criteria:

* Any subject that does not meet the inclusion criteria
* Subject with current severe H. pylori infection
* Subject ingested compounds that may interfere with detection of H. pylori e.g. 4 weeks for all antibiotics, 2 weeks for Bismuth preparations or proton pump inhibitors prior to EGD/collection
* Subject recently tested, less than 3 months and knowledge of H. pylori absence
* Subject tested, less than one year and knowledge of H. pylori presence but NOT undergone prescribed treatment
* Pregnant or lactating
* Inability or unwilling to perform required study procedures
* Subject is unable or unwilling to provide informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing EGD with biopsy for H. pylori diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori Stool Collection | Through Study Completion, an average of 1 year
  In vitro diagnostic (IVD) device performance

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - One (1) Location in Arizonia, Mesa, Arizona
  - One (1) Location in Mission Hills, California, Mission Hills, California
  - One (1) Location in Oxnard, California, Oxnard, California
  - One (1) Location in Florida, Palm Harbor, Florida
  - One (1) Location in Missouri, St Louis, Missouri
  - One (1) Location in Great Neck, New York, Great Neck, New York
  - One (1) Location in North Carolina, Asheville, North Carolina
  - One (1) Location in Ohio, Mentor, Ohio
  - One (1) Location in Greenville, South Carolina, Greenville, South Carolina
  - One (1) Location in Houston, Texas, Houston, Texas
  - One (1) Location in Virginia, Chesapeake, Virginia
- One (1) Location in Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided